CLINICAL TRIAL: NCT05863052
Title: Analyzing Clinical Outcomes and Genomic Data of American Indian Patient Population Treated With Immune Checkpoint Inhibitors for Various Cancers
Brief Title: Analyzing Clinical Outcomes and Genomic Data of American Indian Patient Population
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-ClinO+GenD; BAA PMWP 213 (Other Grant/Funding Number: FDA); OU202111ARN-OKAMERICANINDIAN (Other: OUHSC)
Record Dates: First submitted 2023-03-13; First posted 2023-05-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Immune Checkpoint Inhibitors; Metastatic Solid Tumor; Nonsmall Cell Lung Cancer; Melanoma; Renal Cell Carcinoma; Gastrointestinal Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Gastrointestinal Neoplasms; Carcinoma, Squamous Cell | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- American Indian population
  Interventions: Biological: Immunotherapy
- Caucasians treated with immunotherapy
  Interventions: Biological: Immunotherapy

INTERVENTIONS:
Biological: Immunotherapy — immunotherapy

SUMMARY:
The aim of this study is to describe the outcomes in American Indian patients receiving immunotherapy in a multi-institution retrospective study at several other high-volume centers that care for this patient population and to identify any healthcare disparities that can lead to future interventional studies.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors have been shown to increase survival in metastatic solid tumor patients when compared to the previously standard of care chemotherapy. Epidemiologic studies of American Indian cancer patients demonstrated having significantly worse survival when compared with Caucasians when controlled for age, sex, alcohol abuse, smoking, insurance, and disease stage.

There are no current studies specifically examining the American Indian population receiving treatment with immune checkpoint inhibitors. The aim is to describe the outcomes in American Indian patients receiving immunotherapy in a multi-institution retrospective study at several other high-volume centers that care for this patient population and to identify any healthcare disparities that can lead to future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* above age 18,
* histologically and cytologically confirmed NSCLC, melanoma, head and neck squamous cell carcinoma, gastrointestinal cancers,, renal cell carcinoma, or any other solid tumors where immune checkpoint therapy has been used
* received immunotherapy as part of their treatment
* Self-identified American Indian in ethnicity
* Patients at the Stephenson Cancer Center between 2015 to 2021

Exclusion Criteria:

* patients who did not receive immune checkpoint inhibitor therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: American Indian population is the primary group of interest for this study.
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Evaluating progression free survival of American Indian population vs. White population who were treated with immunotherapy
Overall Survival Benefit | 1 year
  Evaluating the overall survival benefit of American Indian population vs. white population who were treated with immunotherapy
Treatment related Adverse Events | 1 year
  Evaluating treatment related adverse events of American Indian population vs. white population who were treated with immunotherapy

SECONDARY OUTCOMES:
Difference in cancer related mortality | 1 year
  Evaluate the difference in cancer related mortality in American Indian populations vs white

OTHER OUTCOMES:
Tumor mutational burden | 1 year
  Describe the differences in tumor mutational burden (TMB) between the American Indian population vs Whites or Black Americans
Somatic genetic variants | 1 year
  Describe the somatic genetic variants differences between the American Indian population vs Whites or Black Americans
Demographic differences | 1 year
  Describe the demographics differences between the American Indian population vs Whites or Black Americans

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Naqash, MD, Principal Investigator — University of Oklahoma
Locations (6):
- United States (6):
  - Arizona Cancer Center at the Unvieristy of Arizona, Tucson, Arizona
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Monument Health Cancer Care Institute, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No